CLINICAL TRIAL: NCT01195220
Title: Project AWARE: Using the ED to Prevent STIs in Youth
Brief Title: Project AWARE: Using the Emergency Department (ED) to Prevent Sexually Transmitted Infections (STIs) in Youth
Acronym: AWARE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We could not obtain proper funding to complete this study.
Sponsor: North Bronx Healthcare Network (Other)
Responsible Party: Principal Investigator, Yvette Calderon,MD, MS, Director of the Urgent Care Clinic, North Bronx Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010-381
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Chlamydia; Gonorrhea; HIV
Keywords: STI screening; Emergency Department; Chlamydia; Gonorrhea; HIV; behavior; teenagers; intervention
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Emergencies; Behavior | interventions — HIV Testing

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- HIV-T (Active Comparator): Group 1, the control, will be the current standard of care, consenting video and testing for HIV alone (HIV-T).
  This is the current standard of care. It obtains consent for HIV vesting by a proven video, and provides rapid HIV testing on site. Informed consent video includes information about the test and its interpretation, as mandated by New York State Law. The the OraQuick ADVANCE® Rapid HIV- 1/2 Antibody Test
  Interventions: Behavioral: HIV testing
- STI/HIV-T (Experimental): Group 2 will add routine STI testing for CT and GC, (STI/HIV-T).
  This intervention adds testing for GC and CT to HIV testing. The informed consent video will incorporate information for STIs to accompany information presented on HIV. GC and CT screening is conducted via a urine sample. The APTIMA Combo 2 Assay has been cleared by the Food and Drug Administration for sale in the US. It employs Gen-Probe's patented Transcription-Mediated Amplification (TMA) technology to detect CT and GC using urine specimens for both male and female patients. We will test urine for GC and CT at the ED visit using the hospital lab within the urban ED.
  Interventions: Behavioral: STI/HIV-T
- STI/HIV-Plus (Experimental): Group 3, in addition to combined STI/HIV testing, will add a behavioral video encouraging safer sex, which is chosen for participants based on their answers to a brief measure on stage of change (STI/HIV-PLUS).
  This intervention includes the combined STI/HIV testing, and adds the behavioral video that encourages safer sex and is targeted to the participants' stage of change. While patients wait for their HIV test result (20-30 minutes), patients will view these video vignettes
  Interventions: Behavioral: STI/HIV-T; Behavioral: STI/HIV-Plus

INTERVENTIONS:
Behavioral: HIV testing — This is the current standard of care. It obtains consent for HIV vesting by a proven video, and provides rapid HIV testing on site. Informed consent video includes information about the test and its interpretation, as mandated by New York State Law. The the OraQuick ADVANCE® Rapid HIV- 1/2 Antibody Test
  Arms: HIV-T
Behavioral: STI/HIV-T — This intervention adds testing for GC and CT to HIV testing. The informed consent video will incorporate information for STIs to accompany information presented on HIV. GC and CT screening is conducted via a urine sample. The APTIMA Combo 2 Assay has been cleared by the Food and Drug Administration for sale in the US. It employs Gen-Probe's patented Transcription-Mediated Amplification (TMA) technology to detect CT and GC using urine specimens for both male and female patients. We will test urine for GC and CT at the ED visit using the hospital lab within the urban ED.
  Arms: STI/HIV-Plus; STI/HIV-T
Behavioral: STI/HIV-Plus — This intervention includes the combined STI/HIV testing, and adds the behavioral video that encourages safer sex and is targeted to the participants' stage of change. While patients wait for their HIV test result (20-30 minutes), patients will view these video vignettes.
  Arms: STI/HIV-Plus

SUMMARY:
Project Aware introduces a sexually transmitted infection (STI) screening model for sexually experienced adolescents aged 14 to 21 in a large, inner-city Emergency Department (ED) in the Bronx, N.Y. Project Aware will scaffold routine, rapid testing and counseling for Chlamydia trachomatis (CT) and Neisseria gonorrhoeae (GC) onto an existing, successful, ED-based HIV testing and counseling program, Project BRIEF. Project Aware will educate and motivate youth to use condoms with the aid of a theory-based, youth-friendly multimedia behavioral intervention proven to be effective during the investigator's K23 training. Through Project Aware, the investigators propose to change the paradigm of STI testing. Whereas a view of "HIV exceptionalism" has persisted in U.S. health policies on STI testing, the investigators propose a comprehensive approach, in which efforts to identify, treat, and prevent multiple STIs coalesce in one program. The research study has two phases. In the production phase, new STI material will be added to the multimedia intervention currently used for HIV education. In the evaluation phase, a randomized controlled trial (RCT) will be conducted to assess the effectiveness of Project Aware in identifying, treating, and preventing new STI infections among high-risk adolescents. The RCT is designed to test the incremental effectiveness of three STI prevention methods: (1) HIV testing and counseling (T&C), (2) HIV T&C and STI testing, and (3) HIV/STI Testing plus a point-of-service risk reduction video that incorporates both HIV and STI counseling and education. The study is powered to examine three STI prevention outcomes: (1) the number of STI infections identified and treated successfully at baseline; (2) the number of new STI infections over the 12 months following study entry, identified by (a) performing STI testing at each follow-up assessment; and (b) obtaining anonymized rate data on STIs reported to the New York City Department of Health; (3) condom use behavior. 600 youth aged 14-21 will be enrolled in the RCT. Youth will be approached in the ED waiting room and recruited by Public Health Advocates. All will complete a survey to screen for eligibility; eligible youth will complete the baseline measures and be randomized. The follow-up data points and measures will be followed at 4, 8 and 12 months (4 time points) and STI testing will be included.

DETAILED DESCRIPTION:
Almost half of all new sexually transmitted infections (STIs) occur in young people aged 15-24.1 The vast majority (88%) consists of chlamydia (CT), gonorrhea (GC), human papilloma virus (HPV), and trichomoniasis.1 Additionally, the Centers for Disease Control and Prevention (CDC) reported that young people aged 15-24 accounted for 7,297 new HIV diagnoses in 2008, 17.7% of all new diagnoses for the year.2 Inner-city, sexually active adolescents are exceptionally vulnerable to contracting HIV and STIs.3 In 2008, the Bronx had the highest proportion of AIDS cases of any borough in New York City.5 For Bronx females aged 15 to 19, the CT infection case rate was 7,621 per 100,000 and 812 per 100,000 for GC, the highest in this age group in New York City.4 The infection rate among young men aged 15-19 in the Bronx is also the highest in New York City: the case rate was 2,092 for CT and 458 for GC.4

Based on its concern about adolescent HIV risk, the CDC changed the HIV testing paradigm by recommending routine HIV testing for all adolescents. It also recommended routine HIV screening for all patients seeking STI testing and treatment at STI clinics.6 However, universal STI screening in adolescents is not routine in other medical settings, even though most STIs are asymptomatic and therefore undiagnosed. We believe that screening youth for HIV provides an opportunity to screen for STIs as well, and that testing should be combined with harm reduction interventions. This project will evaluate the efficacy of Project AWARE in diagnosing, treating, and preventing HIV and STI infections in a Bronx Emergency Department (ED).

This proposal is based on eight years of research and experience developing and testing a successful ED-based multimedia program for HIV prevention.7 The first four years focused on developing videos that educated adult ED patients and encouraged them to be tested for HIV. Project BRIEF-A has achieved high acceptance (95%) for adult HIV testing and has linked 85% of HIV+ patients into specialized medical care.8,9 The last 4 years developed Project BRIEF-T, an efficient, youth-friendly, theory-based harm reduction video intervention for teens.10 It delivered different short video interventions to youth based on their stage of change. Results are promising: Project BRIEF-T was effective in moving youth to the next stage of change in their intentions to use condoms. We propose in this application to test Project AWARE, which will add universal STI testing to Project BRIEF-T, and evaluate the effects of the theory-based video intervention on condom use at 4, 8, and 12 months post-testing.

Project AWARE will be evaluated using a three group randomized trial. Group 1, the control, will be the current standard of care, consenting video and testing for HIV alone (HIV-T). Group 2 will add routine STI testing for CT and GC, (STI/HIV-T). Group 3, in addition to combined STI/HIV testing, will add a behavioral video encouraging safer sex, which is chosen for participants based on their answers to a brief measure on stage of change (STI/HIV-PLUS). Comparing Group 1 to Group 2 will identify the number of new STI infections identified through routine testing to establish whether routine screening successfully identified a substantial number of new cases over and above routine care. Comparing Group 1 to Group 3 will identify whether the addition of the Stages of Change intervention significantly increases condom use among teens.

Specific Aims:

1. To compare the efficacy of the three study arms and to test for significant differences at the 4 month follow up in order to provide information to programs concerning efficient use of resources.
2. To study the persistence of the intervention effects over time between 4 and 12 months on the primary outcome as well as to examine the intervention effect on condom use intentions, condom self-efficacy, and condom outcome expectancy and reduce sexual risk behavior, at each follow up time point.
3. To estimate the prevalence of STIs at baseline.

The project is explicitly translational. If Project AWARE efficiently identifies and treats asymptomatic HIV and STIs, and successfully reduces subsequent sexual risk behavior among teens, it can be implemented in EDs at relatively low cost. Given the new emphasis in the U.S. on efficient preventive care, this project can provide an exemplary portable intervention tool that can reach many high risk youth with asymptomatic STIs and HIV who do not access routine primary care. The study's results might also contribute to the development of new screening policies to incorporate multiple STIs into existing HIV screening.

ELIGIBILITY:
Inclusion Criteria:

* 14-21 years old
* Sexually active
* English speaking

Exclusion Criteria:

* medically unstable
* unable to understand the consent process
* tested for HIV/STI within the past 4 weeks

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
STI infections (GC and CT) | 4-months post intervention

SECONDARY OUTCOMES:
intentions for condom use | immediately after intervention (baseline)
Intention for condom use | 4-months post intervention
Intention for Condom Use | 8 months post intervention
Intentions for Condom Use | 12 months post intervention
STI infections (GC and CT) | 8-months post intervention
STI infections (GC and CT) | 12 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Calderon, MD, MS, Principal Investigator — Jacobi Medical Center, Albert Einstein College of Medicine
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States